CLINICAL TRIAL: NCT03145727
Title: Transcutaneous Electric Nerve Stimulation Effects on Nausea and Vomit Chemotherapy-induced
Brief Title: Electric Stimulation on Nausea and Vomit Chemotherapy Induced
Acronym: TENS-NV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TENS-NV-2017
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer Female; Acupuncture
Keywords: Chemotherapy; nausea; vomiting; transcutaneous electrical acupoint stimulation
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: The selection of the investigated will be characterized as non-probabilistic with a convenience approach, whose patients will be included in the study sequentially until the necessary sizing has been achieved. Patients will be included sequentially for convenience (according to the inclusion and exclusion criteria) and non-probabilistic. The included individuals will be randomly randomized by Random Allocation System software in three groups, 1) placebo group; 2) High Frequency Group; 3) Low Frequency Group.
Who Masked: Participant
Masking Description: The participant will be blind to the TENS allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Group (Placebo Comparator): Placebo Group: In this group the participants received TENS with frequency of 75Hz, pulse duration of 200 microseconds. The stimulation time will be for only 10s.
  Interventions: Device: Placebo Group
- Low Frequency Group (Experimental): Low Frequency Group: In this group the TENS will be adjusted with frequency of 10Hz, pulse duration of 200 microseconds. The stimulation time will be 30 minutes and the intensity will be constantly adjusted in order to keep as high as possible within the tolerance threshold of the patient.
  Interventions: Device: Low Frequency Group
- High Frequency Group (Experimental): High Frequency Group: In this group the TENS will be adjusted with frequency of 150Hz, pulse duration of 200 microseconds. The stimulation time will be 30 minutes and the intensity will be constantly adjusted in order to keep as high as possible within the tolerance threshold of the patient.
  Interventions: Device: High Frequency Group

INTERVENTIONS:
Device: Placebo Group — In this group, the TENS will be administered by 30 minutes prior to chemotherapy administration with the stander electrodes positions, in the opposite arm of the chemotherapy infusion, but in this group the electrical stimulation will be performed just by 10 seconds and turn off for all reminiscent time of the protocol.
  Arms: Placebo Group
Device: Low Frequency Group — In this group the TENS will be administered by 30 minutes prior to chemotherapy administration with the stander electrodes positions, in the arm opposite the chemotherapy infusion. The electrical stimulation will be continued for all time secession. The electrical pulse parameters will be setting according describe early.
  Arms: Low Frequency Group
Device: High Frequency Group — In this group the TENS will be administered by 30 minutes prior to chemotherapy administration with the stander electrodes positions, in the arm opposite the chemotherapy infusion. The electrical stimulation will be continued for all time secession. The electrical pulse parameters will be setting according describe early.
  Arms: High Frequency Group

SUMMARY:
Chemotherapy induces nausea and vomit for some large patients. But, some chemotherapy protocol has a high indices of the incidence as observed in a combination of Anthracycline and Cyclophosphamide (AC). To prevent this symptoms, some medication can be used as Ondansetron. By other hands, the traditional acupuncture on Chinese Medicine have been used a PC6 point to avoid nausea and vomit. More recently, a transcutaneous electric nerve stimulation (TENS) also has been used for this application. Our study will test the TENS applied on PC6 point with two different frequencies (high and low) to evaluated the nausea and vomit inhibition effects.

DETAILED DESCRIPTION:
We will enroll 84 women that being starts a chemotherapy protocol with a Anthracycline and Cyclophosphamide (AC) as a part of breast cancer treatment. All volunteers will be submitted a 30 minutes TENS prior to chemotherapy administration. Three different TENS treatment will be test: 1) placebo; 2) high frequency and 3) low frequency. The self-adhesive electrodes will be positioned in the same position for all different TENS treatment (opposite arm to the chemotherapy infusion). The eletctrodes will be positioned as follows: the first electrode at the PC6 point which is located proximal to the flexion fold of the wrist in the middle of the anterior face of the forearm, between the tendons of the long palmar and radial flexor muscles of the carpus and the second electrode at any point in the hand. After that, all volunteers will receipt a formulary to self-complete a nausea and vomit symptoms record during the next 24 hours. Number of incidence and magnitude of the symptoms will express the accumulated indices the occurrence and severity of the symptoms, as further describe in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Having breast cancer diagnosed through anatomopathological investigation;
* Indication of neoadjuvant or adjuvant chemotherapy treatment with the combination of anthracycline and cyclophosphamide associated with Ondasetron used as a routine of the Santa Rita Hospital chemotherapy service;
* Present Karnofsky score (KPS) higher than 70 points;
* Being female;
* Be between 18 and 65 years of age and be able to participate in outpatient chemotherapy.

Exclusion Criteria:

* Patients with breast cancer treated with chemotherapeutic regimens other than anthracycline and cyclophosphamide;
* Inability to report nausea and vomiting due to neurological changes, difficulty understanding and / or lack of caregivers that may contribute to the completion of the report;
* Be submitted to radiation therapy concomitant with chemotherapy;
* Presence of gastrointestinal and cerebral metastases;
* Presence of cardiac pacemaker;
* Presence of active skin infection in PC6;
* Nausea and vomiting caused by electrolyte disturbances or intestinal;
* Presence of intra-cranial hypertension.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with indication for neoadjuvant or adjuvant chemotherapy treatment with the combination of anthracycline and cyclophosphamide associated with Ondasetron
Enrollment: 84 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative index of nausea | Cumulative index of nausea in the first 24 hours after an infusion of chemotherapy.
  The 24-hour follow-up record of symptoms of nausea and vomiting will be performed using a form developed from the MASEM anti-emetic instrument (MAT), especially for the present study. This form includes a diary to record emetic events within 24 hours after the administration of chemotherapy. Thus, we will evaluate: the cumulative index of nausea and vomiting over 24 hours after the infusion of the first cycle of high grade emetic chemotherapy.Participants will be instructed to fill out the instrument and take the questionnaire home, bringing it back to the investigators when they return to the outpatient clinic for another round of chemotherapy.

SECONDARY OUTCOMES:
Cumulative index of episodes of vomiting | Cumulative index of episodes of vomiting in the first 24 hours after an infusion of chemotherapy.
  The 24-hour follow-up record of symptoms of nausea and vomiting will be performed using a form developed from the MASEM anti-emetic instrument (MAT), especially for the present study. This form includes a diary to record emetic events within 24 hours after the administration of chemotherapy. Thus, we will evaluate: the cumulative index of nausea and vomiting over 24 hours after the infusion of the first cycle of high grade emetic chemotherapy.Participants will be instructed to fill out the instrument and take the questionnaire home, bringing it back to the investigators when they return to the outpatient clinic for another round of chemotherapy.
Intensity of nausea symptoms | Intensity of the symptom of nausea within the first 24 hours after infusion of chemotherapy.
  As for the intensity of nausea, a Visual Analog Scale will be used to help measure the intensity of each patient. The instrument will question the patient about the degree of nausea and it will provide an auto report with a note that can vary from 0 to 10, with note 0 representing absence of the symptom while note 10 represents the most intense sensation experienced by the patient . Participants will be instructed to fill out the instrument and take the questionnaire home, bringing it back to the investigators when they return to the outpatient clinic for another round of chemotherapy.
Severity of vomiting episodes | Severity of vomiting episodes within the first 24 hours after chemotherapy infusion.
  The severity assessment of vomiting episodes includes a diary to record the number of episodes of vomiting, which may be small, medium or large. Thus, we will assess the severity of vomiting over 24 hours after the infusion of the first cycle of high grade emetic chemotherapy. Participants will be instructed to complete the instrument and take the questionnaire home, bringing it back to the investigators. When they return to the clinic for another round of chemotherapy.
Need for rescue antiemetic | Need for rescue antiemetic within the first 24 hours after chemotherapy infusion
  The 24-hour follow-up record of symptoms of nausea and vomiting will be performed using a form developed from the MASEM anti-emetic instrument (MAT), especially for the present study. This form includes a diary to record emetic events within 24 hours after the administration of chemotherapy. Thus, we will evaluate: the cumulative index of nausea and vomiting over 24 hours after the infusion of the first cycle of emetic high-grade chemotherapy, the volume of vomiting in each episode and the need for rescue antiemetics will also be recorded. Will be instructed to fill out the instrument and take the questionnaire home, bringing it back to the researchers when they return to the clinic for their second course of chemotherapy.
Edmonton Symptom Assessment Scale | At the end of 24 hours, you will be asked to complete the Edmonton Symptom Assessment Scale
  At home and at the end of 24 hours, will be asked to fill in the Edmonton Symptom Assessment Scale where symptoms of pain, tiredness, drowsiness, appetite, nausea, shortness of breath, depression, anxiety and well-being will be evaluated, Based on the Brazilian Consensus on Nausea and Vomiting. It is a scale where the patient provides an auto-report with a note that can vary from 0 to 10, with note 0 representing absence of the symptom while note 10 represents the most intense sensation experienced by the patient.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Fabrício Edler Macagnan, Porto Alegre, Rio Grande do Sul
  - Comitê de Ética em Pesquisa - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No